CLINICAL TRIAL: NCT00544479
Title: Is Routine Chest-X-Ray Necessary After Bronchoscpy With Thransbronchial Biopsie? A Prospective Study
Brief Title: No Routine CXR After Bronchoscopy
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr. G. Izbicki, Head Pulmonary Institute, Shaare Zedek Medical Center
Other Study IDs: 180964CTIL
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Most pulmonologist request a routine chest-x-ray after bronchoscopy with transbronchial biopasie to exclude pneumothorax. We published a study in CHEST showing that routine chest-ray might not be necessary. We would like to conduct a propsective study to validate the results of the CHEST-study. Before and after the procedure follwing information will be collected: Age, Sex, Indication for procedure, number of biopsies and segment of biopsie, Saturation, Physical examination, Symptoms suggestive of pneumothorax. If there is no aggravation of the symptoms and/or physical examination after the procedure, as compared to before, routine chest-x-ray will NOT be done. A phone will be made 24 to 48 hours following the procedure to the patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients with bronchoscopy and transbronchial biopsie

Exclusion Criteria:

* No informed consent given

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with bronchoscopy and transbronchial biopsies will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Izbicki, M.D., Principal Investigator — Shaare Zedel Medical Center
Locations (1):
- Institue of Pulmonology, Shaare Zedek M.C., Jerusalem, Israel

REFERENCES:
- [Result] Izbicki G, Shitrit D, Yarmolovsky A, Bendayan D, Miller G, Fink G, Mazar A, Kramer MR. Is routine chest radiography after transbronchial biopsy necessary?: A prospective study of 350 cases. Chest. 2006 Jun;129(6):1561-4. doi: 10.1378/chest.129.6.1561. PMID 16778275